CLINICAL TRIAL: NCT00003661
Title: A Pilot Study of Unrelated Umbilical Cord Blood Transplantation in Children and Adults With Hematologic Malignancies
Brief Title: Chemotherapy, Radiation Therapy, and Umbilical Cord Blood Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Barbara Bambach, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066754; RPCI-RP-9801 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neuroblastoma
Keywords: recurrent childhood acute lymphoblastic leukemia; stage 4S neuroblastoma; recurrent childhood lymphoblastic lymphoma; recurrent adult acute lymphoblastic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neuroblastoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Antilymphocyte Serum; Busulfan; Cyclosporine; Melphalan; Methylprednisolone; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclosporine
Drug: melphalan
Drug: methylprednisolone
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Umbilical cord blood transplantation may be able to replace cells destroyed by chemotherapy or radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy, radiation therapy, and umbilical cord blood transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rates of hematologic and immune reconstitution in pediatric patients with high risk hematologic malignancies in first remission or in second or subsequent remission, and adult patients with acute lymphocytic leukemia (ALL) or acute nonlymphocytic leukemia (ANLL) in second or subsequent remission, who are undergoing high dose chemoradiotherapy followed by unrelated umbilical cord blood (UCB) transplantation. II. Determine the incidence of graft-versus-host disease in this setting. III. Determine whether contamination of umbilical cord blood with maternal cells is a clinical problem in this setting. IV. Describe the incidence of leukemic relapse in these patients after UCB transplantation. V. Describe the incidence of serious infections and secondary lymphoproliferative diseases following transplantation with UCB in these patients. VI. Determine specifically whether larger recipients (greater than 40 kg) can be durably engrafted with unrelated UCB, and determine whether nucleated cell or progenitor cell content of the graft is predictive of hematological engraftment.

OUTLINE: Patients undergo a back-up bone marrow harvest prior to treatment. Patients receive 9 fractions of total body irradiation (TBI) on days -9 to -5, followed by melphalan IV on days -4 to -2 and antithymocyte globulin IV or methylprednisolone IV on days -3 to -1. If TBI is not allowed, busulfan is substituted and administered orally every 6 hours for 4 days on days -8 to -5. On day 0, patients receive umbilical cord blood infusion. Cyclosporine and methylprednisolone begin on day -2 and continue for 6 months. Patients are followed indefinitely for survival and late toxicity.

PROJECTED ACCRUAL: A minimum of 48 patients will be accrued into this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignancy including: - Pediatric acute lymphocytic leukemia (ALL) in first complete remission with high risk features including presence of t(4;11) or t(9;22), or extreme hyperleukocytosis (initial WBC greater than 500 K/mL), or failure to achieve a complete remission after standard induction therapy - Adult ALL or acute nonlymphoblastic leukemia (ANLL) in first complete remission with t(8;14) translocation or failure to achieve complete remission after standard induction therapy - ALL or ANLL in second or subsequent remission - Chronic myelogenous leukemia in chronic or accelerated phase - Myelodysplastic syndrome with evidence of evolution to acute myeloid leukemia Refractory anemia with excess blasts Refractory anemia with excess blasts in transformation Chronic myelomonocytic leukemia - T-lymphoblastic non-Hodgkin's lymphoma in second or subsequent remission - Stage IV neuroblastoma Must also meet all the following conditions: No HLA-ABC/DR identical related bone marrow or UCB donor No 5/6 antigen matched related bone marrow or UCB donor Condition precludes waiting to search and find a donor in the National Marrow Donor Registry Must have an available serologic matched umbilical cord blood unit in the New York Blood Center's Placental Blood Project No active CNS disease Not eligible for COBLT study (Transplantation of Banked Umbilicial Cord Blood Cells for Use in Clinical Research on Transplantation of Umbilical Cord Blood Stem and Progenitor Cells)

PATIENT CHARACTERISTICS: Age: Under 55 at time of umbilical cord blood transplantation Performance status: Zubrod 0-1 Lansky 80-100% Karnofsky 80-100% Life expectancy: At least 3 months Hematopoietic: Adequate hematologic status at time of back-up bone marrow harvest: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: ALT/AST no greater than 4 times normal Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 50 mL/min Cardiovascular: Normal cardiac function by echocardiogram or radionuclide scan (shortening fraction or ejection fraction at least 80% of normal value for age) Pulmonary: FVC and FEV1 at least 60% of predicted for age For adults: DLCO at least 60% of predicted Other: No active infections at time of back-up bone marrow harvest or pretransplant reduction Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Max Age: 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 1998-06; Primary Completion 1999-11 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jean Bambach, MD, Study Chair — Roswell Park Cancer Institute
Locations (17):
- United States (17):
  - University of Florida Health Science Center, Gainesville, Florida
  - Division of Pediatric Surgery, Jacksonville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - New York Blood Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina School of Medicine, Columbia, South Carolina